CLINICAL TRIAL: NCT06873750
Title: A Pilot Study in Defining the Potential of Transcranial Alternating Current Neuromodulation for Stabilizing Memory and Improving Functional Connectivity in Neurodegeneration
Brief Title: Neuromodulation and FMRI in Neurodegenerative Diseases Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Bojana Stefanovic, Director and Senior Scientist, Physical Sciences, Hurvitz Brain Sciences Research Program, Sunnybrook Research Institute, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5787
Record Dates: First submitted 2023-11-21; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment; Traumatic Brain Injury; Neurodegeneration
Keywords: Transcranial Alternating Current Stimulation; Neuromodulation; Functional Magnetic Resonance Imaging; Cognitive Assessment
MeSH Terms: conditions — Cognitive Dysfunction; Brain Injuries, Traumatic; Nerve Degeneration | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This study will follow a single group assignment model. All participants will receive the tACS treatment. The primary goal is proof-of concept that tACS is a feasible, non-invasive treatment that provides some amelioration in working memory, correlated with observable changes in EEG and fMRI imaging metrics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): All participants will receive transcranial alternating current stimulation.
  Interventions: Device: Transcranial Alternating Current Stimulation

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation — Application of low amplitude alternating electric current across the participant's scalp.
  Other Names: Soterix Medical MxN-33 high definition transcranial electrical stimulator

SUMMARY:
In addition to neuronal loss, dysfunction in brain network connectivity has been identified as a correlate of cognitive deficits in neurodegenerative and post-traumatic brain injury states. Transcranial alternating current stimulation (tACS) has been suggested as a promising, non-invasive, method of normalizing network connectivity and hence improving cognition, notably memory. This study will examine the efficacy of tACS at improving working memory performance in patients with neurodegeneration and its correlation to changes in network connectivity, based on functional magnetic resonance imaging (fMRI) and electroencephalography (EEG) imaging data.

DETAILED DESCRIPTION:
The participants will first be scanned on a 3T MRI system (at Sunnybrook Health Sciences Centre) using a multi-channel receive head coil.

The MRI protocol will comprise a T1-weighted structural scan to provide anatomical information and guide prescription of the geometry of subsequent functional scans and subsequent tACS montage (stimulation electrode geometry). Next, a Chemical Exchange Saturation Transfer (CEST) sequence will be run. CEST is a non-invasive alternative to positron emission tomography (PET) imaging that will allow us to make measurements of cerebral metabolism. Glucosamine will be used as an orally administered contrast agent. The next sequence of the MRI protocol will be the resting state blood-oxygenation level dependent (BOLD) fMRI, examining brain function while the patient is idle (i.e., not performing a specific task). Finally, a pseudo-continuous arterial spin labeling (pCASL)/BOLD fMRI sequence will be acquired during which participant may intermittently hear a variety of sounds and be asked to perform a simple memory task, inducing stimulus/task processing related neuronal activations in the brain. The pCASL sequence uses radiofrequency (RF) fields to magnetically "tag" blood in the carotid arteries, thus allowing estimation of cerebral blood flow.

EEG recordings will be performed after the MRI scan. Participants will have electrodes affixed to their scalp with a water soluble paste. After electrode application, participants will be escorted to a sound-attenuating chamber for testing. The participant will be seated in a comfortable reclining chair. Instructions will be given to the subject and testing started shortly after. Testing procedures will include monitoring brain responses to sounds or during performance of the aforementioned simple memory task. Sounds will be presented at a comfortable listening level though headphones or speakers.

After the initial baseline MRI and EEG have been acquired, participants will receive 20 minutes of tACS. The tACS will be delivered via a high definition-tACS system (Soterix Medical, New York, NY). The system is currently approved by US Federal Law as an investigational device. The system includes a cap with 32 electrodes that can be used to deliver stimulation. The electrodes will be chosen through finite head modelling to best stimulate the occipitoparietal cortex. The intensity of stimulation delivered through each electrode will not exceed 3 mA, as prescribed by the hardware-based safety limits.

The participants will undergo post-tACS imaging, on the first and final days of treatment administration and at a 1-month follow up visit, using the same sequences as in the baseline scans described above.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 25 years of age;
2. Have no contraindications to MRI
3. Have received 8 or more years of formal education
4. Be fluent in English
5. Cohort a. must be followed at Sunnybrook Health Sciences Center

Cohort a:

* Have been diagnosed with a suspected neurodegenerative disorder or traumatic brain injury (TBI) with memory deficits impacting functional status
* In case of TBI, cognitive impairment has persisted at least three months post-injury
* Received score of 16 or lower on the Mini Mental State Examination (MMSE)

Cohort b:

* Have no prior diagnosis of a neurodegenerative disorder or post-traumatic brain injury cognitive deficits
* Be experiencing healthy aging and be age and sex matched to Cohort a.

Exclusion Criteria:

1. Have any contraindications to MRI
2. Be pregnancy
3. Have any major comorbid medical conditions (as determined by investigators - e.g., comorbid neurological diseases, uncontrolled hypertension or diabetes, malignancy) or major comorbid psychiatric conditions (as determined by investigators - e.g., schizophrenia or bipolar disorder)

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of cognitive benefits post tACS intervention | 2 years
  The first projected outcome is to demonstrate the feasibility of using tACS as a treatment for working memory deficits in patients in neurodegenerative disorders or post-traumatic brain injury cognitive impairment. The success of which will be assessed using the results of neurophysiological testing such as Alzheimer's Disease Assessment Scale-Cognitive (ADAS-cog) scores (with a lower score compared to pre-tACS baseline indicating improved cognition; scale ranges from 0-70 with 0 indicating no cognitive impairment and scores >18 indicating some degree of impairment) and examining if the scores improve before and after administration of tACS.

SECONDARY OUTCOMES:
Use of resting state fMRI functional connectivity to assess acute and lasting neurophysiological effects of tACS | 2 years
  The secondary objective is to assess if the anticipated tACS mediated cognitive improvements are correlated with a neuroimaging metric such as changes in resting state fMRI connectivity.

IPD SHARING:
Plan to Share IPD: No